CLINICAL TRIAL: NCT01515579
Title: A Randomized, Double-blind, Single-centre, Two-period, Cross-over Trial in Healthy Subjects Investigating the Bioequivalence Between the Phase 2 Formulation of Liraglutide at pH 7.7 (Formulation 3) and the Phase 3 Formulation at pH 8.15 (Formulation 4)
Brief Title: Comparison of Two Liraglutide Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1693; 2005-005948-68 (EudraCT Number)
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation 3 (Experimental)
  Interventions: Drug: liraglutide
- Formulation 4 (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — One single dose of 6.25 mg/mL administered subcutaneously
  Arms: Formulation 3
Drug: liraglutide — One single dose of 6.0 mg/mL administered subcutaneously
  Arms: Formulation 4

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to test for bioequivalence of the phase 3a formulation of liraglutide at pH 8.15 (formulation 4) and liraglutide at pH 7.7 (formulation 3).

ELIGIBILITY:
Inclusion Criteria:

* Good general health as judged by the investigator, based on medical history, physical examination including 12-lead ECG (electrocardiogram), vital signs and blood and urinary laboratory assessments
* BMI (Body Mass Index) of 18.0-27.0 kg/m^2, both inclusive

Exclusion Criteria:

* History of any clinically significant renal, hepatic, cardiovascular, pulmonary, gastrointestinal, metabolic, endocrine, haematological, neurological, psychiatric disease or other major disorders that may interfere with the objectives of the trial, as judged by the Investigator
* Impaired renal function
* Any clinically significant abnormal ECG, as judged by the Investigator
* Active hepatitis B and/or active hepatitis C
* Positive human immunodeficiency virus (HIV) antibodies
* Known or suspected allergy to trial product(s) or related products
* Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures
* Use of any prescription or non-prescription medication, except for paracetamol and vitamins, as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2006-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve (0-t)
Cmax, maximum concentration

SECONDARY OUTCOMES:
Area under the curve
tmax, time to reach Cmax
t½, terminal half-life
Terminal elimination rate constant
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Lund, Sweden

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com